CLINICAL TRIAL: NCT05906290
Title: Formative Development of a Multigenerational eHealth Intervention for Grandparents and Grandchildren
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Stopped Early Due to COVID Restrictions
Sponsor: University of Miami (Other)
Collaborators: Center on Aging and Adult Development Disabilities (CADD) (Unknown)
Responsible Party: Principal Investigator, Sara StGeorge, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20171095
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multigenerational eHealth Intervention for Grandparents and Grandchildren Group (Experimental): Participants in this group will have access to eHealth intervention for 2 weeks.
  Interventions: Other: Multigenerational eHealth Intervention for Grandparents and Grandchildren

INTERVENTIONS:
Other: Multigenerational eHealth Intervention for Grandparents and Grandchildren — Participants in this group will use an online program for 30-45 minutes per week over the course of 2 weeks delivered via smartphone, focusing on increasing physical activity.

SUMMARY:
This study develops a multigenerational electronic Health (eHealth) (web and mobile phone-based) program to improve physical activity levels and to better understand the relationship between grandparents and their grandchildren. The importance of social and familial support for older adults and the need to address increasing declines in physical activity for both children and older adults. Health promotion interventions that capitalize on the existing relationship between grandparents and grandchildren may simultaneously improve health-related outcomes for older adults and children.

ELIGIBILITY:
Inclusion Criteria:

* Female or male grandparent with a grandchild
* Grandparent is at least 45 years old
* Grandparent has a grandchild between the ages of 6-12 years old
* Grandparent is English or Spanish speaking

Exclusion Criteria:

* Grandparent has a chronic medical condition that interferes with physical activity (e.g., wheelchair bound, severe heart disease, uncontrolled hypertension, brittle diabetes mellitus, chronic arthritis)
* Grandparent has a diagnosis of dementia or significant cognitive impairment based on the telephone interview for cognitive status (TICS)

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Program acceptability as measured by Qualitative Interview Guide Field Trial | 2 weeks
  Program acceptability will be measured by Qualitative Interview Guide Field Trial. Participants indicate whether they like the program in a qualitative exit interview. The interview guide consists of 13 open-ended questions regarding the participant's experience testing the program. Acceptability will be based on emergent themes.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M St. George, PhD, Principal Investigator — University of Miami

REFERENCES:
- [Result] Kobayashi MA, St George SM, Leite RO, Noriega Esquives B, Wetstone R, Pulgaron ER, Prado G, Czaja SJ. Formative Development of a Technology-Based Physical Activity Intervention for Grandparents and Grandchildren. J Aging Phys Act. 2022 Jun 1;30(3):482-494. doi: 10.1123/japa.2020-0481. Epub 2021 Oct 5. PMID 34611054